CLINICAL TRIAL: NCT06119282
Title: The Effect of Aromatherapy on Acute Pain Anxiety and Comfort Levels in Women With Primiparous Cesarean Section Randomized Controlled Study
Brief Title: The Effect of Aromatherapy in Women With Primiparous Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gülnihal ARTUĞ CANSIZLAR, MSc. Gynecology and Obstetrics Nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: The Effect of Aromatherapy
Record Dates: First submitted 2022-12-22; First posted 2023-11-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aromatherapy; Cesarean Section Complications; Primiparity; Postpartum Period
Keywords: Aromatherapy; Cesarean Section; Primiparity; Postpartum Period
MeSH Terms: interventions — Nebulizers and Vaporizers; Control Groups; Massage

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a randomized controlled intervention study to evaluate and compare the effects of massage and inhaler aromatherapy on acute pain, comfort level and anxiety in primiparous cesarean section women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test İnhaler (Experimental): After the cesarean section, at the 8th hour postpartum, the VAS/GCA is evaluated, 4 drops of carrier oil are dropped on the upper and lower parts of the wick of the aroma stick, and then 15-20 drops of the prepared essential mixture are dropped and the woman is explained about its use. By the 8th hour of the postop, 4*1 women are allowed to sniff. Before the application, the 30th and 60th minutes VAS/GOC, vital parameters are evaluated.
  Interventions: Other: inhaler
- Test Massage (Experimental): When the studies conducted with the massage method are examined, back massage is applied for 10-30 minutes. Considering the working conditions of the institution, it is thought that a 10-minute massage may be sufficient for the application. The massage application is started at the postpartum 8th hour and applied for 10 minutes on the postoperative 0th day 1*1, 2 times on the postoperative 1st and 2nd days when the woman feels ready. 30 and 60 minutes before application. then VAS/GCS, vital parameters are monitored.
  Interventions: Other: massage
- Control Group (Active Comparator): Pregnant women included in the control group will be left to clinical care, and pain and vital parameters will be monitored starting from the 8th postoperative hour. The scales applied to the experimental groups will be applied on the 2nd postoperative day. Women in the control group who completed the study will be informed about the postpartum use of aromatherapy. Women who want aromatherapy application will be directed to GETAT center.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: inhaler — Experimental: After the cesarean section, at the 8th hour postpartum, the VAS/GCA is evaluated, 4 drops of carrier oil are dropped on the upper and lower parts of the wick of the aroma stick, and then 15-20 drops of the prepared essential mixture are dropped and the woman is explained about its use. By the 8th hour of the postop, 4*1 women are allowed to sniff. Before the application, the 30th and 60th minutes VAS/GOC, vital parameters are evaluated.
  Arms: Test İnhaler
Other: Control Group — Control Group Pregnant women included in the control group will be left to clinical care, and pain and vital parameters will be monitored starting from the 8th postoperative hour. The scales applied to the experimental groups will be applied on the 2nd postoperative day. Women in the control group who completed the study will be informed about the postpartum use of aromatherapy. Women who want aromatherapy application will be directed to GETAT center.
  Arms: Control Group
Other: massage — Experimental: Test Massage When the studies conducted with the massage method are examined, back massage is applied for 10-30 minutes. Considering the working conditions of the institution, it is thought that a 10-minute massage may be sufficient for the application. The massage application is started at the postpartum 8th hour and applied for 10 minutes on the postoperative 0th day 1*1, 2 times on the postoperative 1st and 2nd days when the woman feels ready. 30 and 60 minutes before application. then VAS/GCS, vital parameters are monitored.
  Arms: Test Massage

SUMMARY:
This study was organized as a randomized controlled trial. The sample was calculated as 120 (Control: 60, Experiment 1:30 Experiment 2:30). Primiparous cesarean section women will be evaluated for pain, postpartum comfort and anxiety levels by using lavender oil, tangerine oil and vetiver oil. The first group will be given inhaler application, the second group will be massage and aromatherapy application. The third group will be the control group.

DETAILED DESCRIPTION:
1. Essential Oils and Preparation Steps:

   Obstetrics and Gynecology Specialist, who has a Phytotherapy Certificate approved by the Ministry of Health, in the selection of essential oils, the creation and dilution of the essential mixture. Instructor Consultancy was received from its member Ayşe Şeyma Küçükakça.
2. Preparation of Essential Mixture:

   It should be preferred to use essential oils as a mixture rather than using them alone. The reason for this is to benefit from the synergy created by essential oils. While a mixture of 5 essential oils is preferred in general use, a maximum of 3 essential oils are used after delivery. Note system is used to create synergy between essential oils. The mixture is created by choosing 1 oil from the top note, middle note and bottom note oils. In the essential blend, the first to be smelled is the top note, the middle note is followed by the top note, and the last is the bottom note. The effect of the oils in the mixture is revealed by the heat, and the effect of the oils in the bottom note is revealed. While creating the essential mixture, essential oils with the same effect are preferred to support the desired effect, and top notes can be used to lighten the aroma of these two oils.

   Mandarin (Citrus Nobilis): Top note is citrus essential oil. It has antimicrobial, antiseptic, antispasmodic, anti-inflammatory, diuretic, sleep quality-enhancing, antidepressant, anxiety and stress relieving properties. There is no known side effects. However, exposure to sunlight should be avoided until 12 hours after the application. It can be used with 3%-50% dilution. It creates synergy with lavender and vetiver.

   Lavender (Lavandula Angustifolia): Middle note is a floral essential oil. Its effects are analgesic, supportive of skin health, antibacterial, anti-inflammatory, antiseptic, relaxant, antipyretic, improving sleep quality, balancing blood pressure, antidepressant, reducing stress, fear and anxiety, and helps panic attacks. There is no known side effects. It can be used in 5%-pure form. Vetiver creates synergy with Mandarin.

   Vetiver (Vetiveria zizanoides): Vetiver is woody essential oil from the base notes. Its effects are analgesic, antibacterial, antimicrobial, helping cell regeneration, antispasmodic, improving sleep quality, reducing anxiety and stress, increasing focus and concentration, antidepressant, helping anger control and helping to get rid of negative emotions such as fear. There is no known side effects. It can be used with 5%-50% dilution. It creates synergy with lavender and tangerine.

   Grape Seed Oil: It is a carrier oil suitable for all skin types. It is antiallergic. It has skin moisturizing properties. It is odorless, tasteless and easily absorbed. It has antioxidant properties. It contains high amount of vitamin E. It helps wound healing and cell regeneration. It has anti-inflammatory and calming properties.
3. Dilution of Essential Oils:

   Essential oils should be diluted with carrier oils. The dilution rate is recommen*ded as 1% for children and 2% for adults. The base oil to be used in dilution is 1% dilution rate as 3 drops of essential oil per 5 ml of base oil. The essential oils to be used in the research will be applied by diluting 1% in order to be easy to tolerate and to reduce the possibility of reaction. 3 drops of tangerine, 2 drops of lavender and 1 drop of vetiver will be added to 10 ml of grape seed oil. As tangerine is the top note, its volatility is high. Therefore, 3 drops will be used. Lavender is the middle note essential oil and again volatile. 2 drops will be added to the essential mixture. Vetiver is a base oil. It is more permanent. Therefore, 1 drop will be used.
4. Inhaler Administration Guide:

   After the cesarean section, at the 8th hour postpartum, the VAS/GCA is evaluated, 4 drops of carrier oil are dropped on the upper and lower parts of the wick of the aroma stick, and then 15-20 drops of the prepared essential mixture are dropped and the woman is explained about its use. By the 8th hour of the postop, 4*1 women are allowed to sniff. Before the application, the 30th and 60th minutes VAS/GOC, vital parameters are evaluated.
5. Massage Application Guide:

   When the studies conducted with the massage method are examined, back massage is applied for 10-30 minutes. Considering the working conditions of the institution, it is thought that a 10-minute massage may be sufficient for the application. The massage application is started at the postpartum 8th hour and applied for 10 minutes on the postoperative 0th day 1*1, 2 times on the postoperative 1st and 2nd days when the woman feels ready. 30 and 60 minutes before application. then VAS/GCS, vital parameters are monitored.

   Before the Application; A room with an average temperature of 25 °C and far from noise is arranged for the massage. An examination table, chair or patient bed of appropriate width (60-65 cm) and height (70-80 cm) is used for the procedure.

   After the postpartum woman is brought to a comfortable position, she is given a side lying/inverted sitting position on the chair and the abdominal region is supported.

   The patient's clothing is removed from his shoulders to the sacral region, exposing his back. If the patient's body is damp and sweaty, it is wiped with a paper towel.

   Hands are washed and warmed by rubbing against each other. According to the patient's back area, 2-4 ml of essential oil, which has been approximately warmed by the bain-marie method, is taken into the palm of the hand and applied to the patient's back and massaged.

   Massage begins in the direction of the heart and by following the direction of the muscle fibers.
6. Control Group Follow-up Guide:

Pregnant women included in the control group will be left to clinical care, and pain and vital parameters will be monitored starting from the 8th postoperative hour. The scales applied to the experimental groups will be applied on the 2nd postoperative day. Women in the control group who completed the study will be informed about the postpartum use of aromatherapy. Women who want aromatherapy application will be directed to GETAT center.

ELIGIBILITY:
Inclusion Criteria

* Being able to speak, read and write Turkish,
* Agree to work with selected essential oils,
* Over 18 years of age and volunteering to participate in the study,
* Being nulliparous
* Not having a previous surgical operation history,
* Not to be a risky pregnancy (HT, Gestational diabetes, asthma, etc.),
* No emergency cesarean section complication (EDT, pregnant with bleeding, etc.),
* Not allergic to aromatherapy oils to be applied,
* Presence of sense of smell.

Exclusion Criteria:

* Wanting to stop working
* Complications during/after cesarean section,
* Being multiparous

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Being able to speak, read and write Turkish, Agree to work with selected essential oils, Over 18 years of age and volunteering to participate in the study, Being nulliparous Not having a previous surgical operation history, Not to be a risky pregnancy (HT, Gestational diabetes, asthma, etc.), No emergency cesarean section complication (EDT, pregnant with bleeding, etc.), Not allergic to aromatherapy oils to be applied, Presence of sense of smell.
Enrollment: 120 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 2 days
  Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end.
  The patient marks on the line the point that they feel represents their perception of their current state. Min: 0, Max: 10
State-Trait Anxiety Inventory | 2 days
  Spielberger, like Raymond Cattell and others before him, made the conceptual distinction between chronic or trait anxiety (a general propensity to be anxious) and temporary or state anxiety (a temporary state varying in intensity). min.: 20- max.: 80
Postpartum Comfort Questionnaire (PPCQ) | 2 days
  İt is decided that the developed PPCQ is a clinically reliable instrument to measure the postpartum comfort of the mothers who give birth. min: 34, Max: 170

CONTACTS AND LOCATIONS:
Overall Officials: Gülnihal ARTUĞ CANSIZLAR, 1, Principal Investigator — Istanbul University Cerrahpasa Florence Nightingale Faculty of Nursing
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Aydin Yildirim T, Kitis Y. The Effect of Aromatherapy Application on Cognitive Functions and Daytime Sleepiness in Older Adults Living in a Nursing Home. Holist Nurs Pract. 2020 Mar/Apr;34(2):83-90. doi: 10.1097/HNP.0000000000000371. PMID 32049695
- [Background] Hajibagheri A, Babaii A, Adib-Hajbaghery M. Effect of Rosa damascene aromatherapy on sleep quality in cardiac patients: a randomized controlled trial. Complement Ther Clin Pract. 2014 Aug;20(3):159-63. doi: 10.1016/j.ctcp.2014.05.001. Epub 2014 May 14. PMID 25129884
- [Background] Ueki S, Niinomi K, Takashima Y, Kimura R, Komai K, Murakami K, Fujiwara C. Effectiveness of aromatherapy in decreasing maternal anxiety for a sick child undergoing infusion in a paediatric clinic. Complement Ther Med. 2014 Dec;22(6):1019-26. doi: 10.1016/j.ctim.2014.09.004. Epub 2014 Sep 30. PMID 25453522
- [Background] Johnson K, West T, Diana S, Todd J, Haynes B, Bernhardt J, Johnson R. Use of aromatherapy to promote a therapeutic nurse environment. Intensive Crit Care Nurs. 2017 Jun;40:18-25. doi: 10.1016/j.iccn.2017.01.006. Epub 2017 Feb 23. PMID 28237089
- [Background] Cankaya S, Ratwisch G. The Effect of Reflexology on Lactation and Postpartum Comfort in Caesarean-Delivery Primiparous Mothers: A Randomized Controlled Study. Int J Nurs Pract. 2020 Jun;26(3):e12824. doi: 10.1111/ijn.12824. Epub 2020 Feb 20. PMID 32078754
- [Background] Keshavarz Afshar M, Behboodi Moghadam Z, Taghizadeh Z, Bekhradi R, Montazeri A, Mokhtari P. Lavender fragrance essential oil and the quality of sleep in postpartum women. Iran Red Crescent Med J. 2015 Apr 25;17(4):e25880. doi: 10.5812/ircmj.17(4)2015.25880. eCollection 2015 Apr. PMID 26023343
- [Background] Einion A. Aromatherapy in midwifery practice. Pract Midwife. 2016 May;19(5):12, 14-5. PMID 27295753
- [Background] Cutshall SM, Wentworth LJ, Engen D, Sundt TM, Kelly RF, Bauer BA. Effect of massage therapy on pain, anxiety, and tension in cardiac surgical patients: a pilot study. Complement Ther Clin Pract. 2010 May;16(2):92-5. doi: 10.1016/j.ctcp.2009.10.006. Epub 2009 Nov 14. PMID 20347840
- [Background] Lee HJ, Ko YL. Back massage intervention for relieving lower back pain in puerperal women: A randomized control trial study. Int J Nurs Pract. 2015 May;21 Suppl 2:32-7. doi: 10.1111/ijn.12299. PMID 26125572
- [Background] Ovayolu Ö. Kemoterapi alan meme kanserli kadınlara uygulanan aromaterapinin semptomlara ve yaşam kalitesine etkisi, Erciyes Üniversitesi Sağlık Bilimleri Enstitüsü Hemşirelik Anabilim Dalı. Doktora Tezi. 2011; Kayseri.3.
- [Background] Özdemir H, Öztunç G. Hemşirelik uygulamalarında aromaterapi. Türkiye Klinikleri Hemşirelik Bilimleri Dergisi. 2013;5(2):98-104.
- [Background] Bilgiç Ş. Hemşirelikte Holistik Bir Uygulama; Aromaterapi. Namık Kemal Tıp Dergisi, 2017; 5(3): 134-141.
- [Background] Kavurmacı M, Tan M. Üremik kaşıntı ve aromaterapi uygulaması. Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi. 2014;3(1):674-82.
- [Background] Zor M, Küçükkelepçe Şimşek D, Gölbaşı Z. Türkiye'de aromaterapinin etkisine yönelik yapılan hemşirelik tezlerinin incelenmesi. Türk J. Clin. Lab. 2021; 1: 77-94.
- [Background] Şimşek Elmalı H, Alpar Ecevit Ş. Sezaryen Sonrası Ağrı ve Hemşirelik Bakımı. IGUSABDER, 2020: 11; 267-278.
- [Background] Çapık A, Özkan H, Ejder Apay S. Loğusaların doğum sonu konfor düzeyleri ve etkileyen faktörlerin belirlenmesi. Dokuz Eylül Üniversitesi Hemşirelik Yüksekokulu Elektronik Dergisi. 2014;7(3):186-192.
- [Background] Karaman Özlü Z, Soydan S, Çapık A, ve ark. Sezaryen ameliyatı olan lohusalarda progresif gevşeme egzersizlerini ağrı kontrolü üzerine etkisi. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi.2016;19(1):58-64.
- [Background] Boz İ, Selvi N. Doğum Sonu Dönemde İyi Bakım Uygulamaları: Kanıtlarla Tamamlayıcı Terapiler. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 2016;19: 25-32.
- [Background] Şahin N, Aydın D, Akay B. Hemşirelik Öğrencilerinin Bütüncül Tamamlayıcı Ve Alternatif Tıbba Karşı Tutumlarının Değerlendirilmesi. Balıkesir Sağlık Bilimleri Dergisi, 2019; 8(1):21-26.
- [Background] Kaufmann C. Aromatic Alchemy For Well-Being. New York; The Country Man Press, 2018.
- [Background] Rathfısch G. Kadın Sağlığında Klinik Aromaterapi. Adana; Çukurova Nobel Tıp, 2019.
- [Background] Ayik C. Ameliyat Öncesi Dönemde Aromaterapi Masajının Anksiyete Ve Uyku Kalitesine Etkisinin İncelenmesi (Yüksek Lisans Tezi). Dokuz Eylül Üniversitesi Sağlık Bilimleri Enstitüsü, 2016.
- See also: Is it safe to use essential oil "neat" (undiluted) on the skin? — http://www.alliance-aromatherapists.org/aromatherapy-safety
- See also: Knowing how to calculate dilutions is crucial to the safe practice of aromatherapy. — http://www.tisserandinstitute.org/essential-oil-dilution-chart/